CLINICAL TRIAL: NCT03254394
Title: Intravenous Lidocaine for Preventing Painful Oxaliplatin-induced Peripheral Neuropathy (OIPN)
Brief Title: Lidocaine for Oxaliplatin-induced Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Assistant Professor of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201705166
Record Dates: First submitted 2017-08-09; First posted 2017-08-18 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Neuropathy, Painful; Chemotherapy-induced Peripheral Neuropathy; Colorectal Cancer
Keywords: Oxaliplatin; Cold hypersensitivity; Neuropathy; Colorectal cancer; CIPN; Neuropathic Pain
MeSH Terms: conditions — Neuropathy, Painful; Colorectal Neoplasms; Cold Hypersensitivity; Neuralgia | interventions — Lidocaine; Folfox protocol

STUDY DESIGN:
Intervention Model Description: Tolerability phase: prospective, open-label Efficacy pilot study: randomized, parallel, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At enrollment, each patient will be assigned a study number, which will match a previously prepared computer-generated list of randomization numbers to determine the interventions. The participants and all other study personnel will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo + FOLFOX (Placebo Comparator): Intravenous infusion of D5W solution over a 130 minute period.
  FOLFOX:
  Oxaliplatin 85mg/m2 IV over 2h, Leucovorin 400 mg/m2 IV over 2h, 5-FU 400mg/m2 IV bolus, followed by a 1200mg/m2/day continuous infusion for 2 days.
  Interventions: Drug: Placebo; Drug: FOLFOX regimen
- Lidocaine + FOLFOX (Active Comparator): Intravenous infusion of lidocaine hydrochloride solution in D5W over a 130 minute period.
  FOLFOX:
  Oxaliplatin 85mg/m2 IV over 2h, Leucovorin 400 mg/m2 IV over 2h, 5-FU 400mg/m2 IV bolus, followed by a 1200mg/m2/day continuous infusion for 2 days.
  Interventions: Drug: Lidocaine Hydrochloride; Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — Intravenous lidocaine will be dosed as a brief 1 mg/kg infusion (based on Ideal Body Weight (IBW)) over 10 minutes, followed by a 0.04 mg/kg/min infusion over additional 120 minutes, resulting in a total dose of 5.8 mg/kg IBW.
  If this dose is tolerable in four consecutive sessions of mFOLFOX6 in six or more of the eight patients in the tolerability phase, we will initiate the randomized efficacy pilot study.
  Arms: Lidocaine + FOLFOX
Drug: Placebo — Dextrose 5% in water will be administered as active comparator.
  Arms: Placebo + FOLFOX
Drug: FOLFOX regimen — Each cycle (repeated every 14 days):
  Oxaliplatin 85mg/m2 IV over 2h, Leucovorin 400 mg/m2 IV over 2h, 5-FU 400mg/m2 IV bolus, followed by a 1200mg/m2/day continuous infusion for 2 days.
  Other Names: mFOLFOX6

SUMMARY:
Oxaliplatin-induced neuropathy is a major dose-limiting side effect in patients with colorectal cancer treated with the FOLFOX chemotherapy regimen. Hypersensitivity to cold is the sensory hallmark of oxaliplatin-induced neuropathy, and it can predict the development of long-term neuropathy. In this study, the investigators aim to determine whether intravenous lidocaine can prevent oxaliplatin-induced cold hypersensitivity.

DETAILED DESCRIPTION:
Colorectal cancer is the third leading cause of cancer death in the United States, with an estimated incidence of 130.000 cases per year. Oxaliplatin is the first-line chemotherapy regimen for gastro-intestinal cancers. Despite its efficacy, oxaliplatin causes peripheral neuropathy in 72% of the treated patients. Acute oxaliplatin-induced peripheral neuropathy [OIPN] is the most common dose-limiting side effect of oxaliplatin and characterized by profound cold allodynia in the extremities. In about 21% of the patients acute OIPN exacerbates into chronic neuropathic pain, which is treatment resistant to currently approved drugs, pointing towards a great need to identify an effective strategy in preventing OIPN. Recent literature suggests that certain methods of assessing sensory nerve function in neuropathic pain patients may provide a prediction to an individual analgesic response; however, no placebo-controlled studies have been performed with the primary goal of identifying treatment response predictors in preventing OIPN.

In this pilot study we will both determine the tolerability and the efficacy of intravenous Lidocaine, for preventing oxaliplatin-induced cold hypersensitivity in the setting of mFOLFOX6 chemotherapy for advanced colorectal cancer.

The proposed study will be conducted in two phases. The tolerability phase is an open-label study to determine the tolerable dose regimen of IV lidocaine in patients with advanced colorectal cancer receiving oxaliplatin chemotherapy. The efficacy pilot phase is a randomized, double-blinded, controlled study comparing the outcomes between IV lidocaine versus placebo in the same setting of colorectal cancer. Consented subjects will attend a screening visit and six intervention visits, during which they will undergo sensory testing and receive intravenous lidocaine or placebo infusion. Cold hypersensitivity and spontaneous pain will be assessed at baseline, daily for 12 weeks and at follow-up visits. At enrollment, each patient will be assigned a study number, which will match a previously prepared computer-generated list of randomization numbers to determine the interventions lidocaine or placebo. The participants and all other study personnel will be blinded to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Stage III and IV colorectal cancer.
* Scheduled for oxaliplatin treatment in mFOLFOX6-based chemotherapy regimen.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Renal insufficiency (defined as calculated Creatinine clearance < 30mL/min)
* Moderate to severe liver failure (defined as ALT or AST > 3 times upper limit of normal if no liver metastases are present; ALT or AST > 5 times upper limit of normal if liver metastases are present).
* Presence of brain metastases.
* Patients with currently uncontrolled cardiac arrhythmias (non-sinus rhythm).
* Patients with history of arrhythmias under pharmacological/pacemaker control will be allowed, except if receiving antiarrhythmic medication listed in "contra-indicated medications".
* Contraindication or allergy to intravenous lidocaine.
* Pre-existing symmetric peripheral painful neuropathy.
* Treated with chemotherapy within the past 12 months.
* Pregnancy or breastfeeding
* Currently treated with any of the following contraindicated medications: Saquinavir, Lopinavir, Amprenavir, Atazanavir, Delavirdine, Mexiletine (and other types of sodium-channel blocker antiarrhythmics), Phenytoin, Carbamazepine, Oxcarbazepine, Lamotrigine, Amiodarone, Dronedarone, Dihydroergotamine, Cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared 6 months after publication of the results in a peer-reviewed journal, upon submission of a robust data analysis plan to the study investigators.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: IPD will be shared 6 months after publication of the results in a peer-reviewed journal, upon submission of a robust data analysis plan to the study investigators.

REFERENCES:
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Attal N, Rouaud J, Brasseur L, Chauvin M, Bouhassira D. Systemic lidocaine in pain due to peripheral nerve injury and predictors of response. Neurology. 2004 Jan 27;62(2):218-25. doi: 10.1212/01.wnl.0000103237.62009.77. PMID 14745057
- [Background] Attal N, Gaude V, Brasseur L, Dupuy M, Guirimand F, Parker F, Bouhassira D. Intravenous lidocaine in central pain: a double-blind, placebo-controlled, psychophysical study. Neurology. 2000 Feb 8;54(3):564-74. doi: 10.1212/wnl.54.3.564. PMID 10680784
- [Result] Ventzel L, Madsen CS, Jensen AB, Jensen AR, Jensen TS, Finnerup NB. Assessment of acute oxaliplatin-induced cold allodynia: a pilot study. Acta Neurol Scand. 2016 Feb;133(2):152-155. doi: 10.1111/ane.12443. Epub 2015 Jun 2. PMID 26032776

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + FOLFOX: Intravenous infusion of D5W solution over a 130 minute period.
  FOLFOX:
  Oxaliplatin 85mg/m2 IV over 2h, Leucovorin 400 mg/m2 IV over 2h, 5-FU 400mg/m2 IV bolus, followed by a 1200mg/m2/day continuous infusion for 2 days.
  Placebo: Dextrose 5% in water will be administered as active comparator.
  FOLFOX regimen: Each cycle (repeated every 14 days):
  Oxaliplatin 85mg/m2 IV over 2h, Leucovorin 400 mg/m2 IV over 2h, 5-FU 400mg/m2 IV bolus, followed by a 1200mg/m2/day continuous infusion for 2 days.
- Lidocaine + FOLFOX: Intravenous infusion of lidocaine hydrochloride solution in D5W over a 130 minute period.
  FOLFOX:
  Oxaliplatin 85mg/m2 IV over 2h, Leucovorin 400 mg/m2 IV over 2h, 5-FU 400mg/m2 IV bolus, followed by a 1200mg/m2/day continuous infusion for 2 days.
  Lidocaine Hydrochloride: Intravenous lidocaine will be dosed as a brief 1 mg/kg infusion (based on Ideal Body Weight (IBW)) over 10 minutes, followed by a 0.04 mg/kg/min infusion over additional 120 minutes, resulting in a total dose of 5.8 mg/kg IBW.
  If this dose is tolerable in four consecutive sessions of mFOLFOX6 in six or more of the eight patients in the tolerability phase, we will initiate the randomized efficacy pilot study.
  FOLFOX regimen: Each cycle (repeated every 14 days):
  Oxaliplatin 85mg/m2 IV over 2h, Leucovorin 400 mg/m2 IV over 2h, 5-FU 400mg/m2 IV bolus, followed by a 1200mg/m2/day continuous infusion for 2 days.
Period: Overall Study
Arm/Group | Placebo + FOLFOX | Lidocaine + FOLFOX
Started | 12 | 14
Completed | 12 | 12
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: This includes only patients who are enrolled and randomized into 2 groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + FOLFOX | Lidocaine + FOLFOX | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (16.4) | 50.9 (13.2) | 51.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Intensity of Oxaliplatin-induced Cold Pain/Unpleasantness vs Time
Description: The intensity of cold pain and cold unpleasantness is evaluated separately, assessed daily on a 0-10 scale, upon holding a pre-cooled (~8°C) metal cylinder for 10 seconds. the area under the curve of cold pain and cold unpleasantness vs time is calculated per chemotherapy cycle (every two weeks) and serves as a primary outcome measure.
  For intervention (lidocaine+FOLFOX) and control (placebo+FOLFOX) groups, the average of cold pain AUC and cold unpleasantness AUC over 7 cycles was calculated. The average AUCs over 7 cycles were compared between study arms.
  The AUC is measured as a score on a 0-10 scale multiplied by 14 days and may range between 0 and 140. Higher AUC values represent more intense cold pain/unpleasantness.
Time Frame: 14 weeks
Population: data for 14 days following the 6th cycle was collected and analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale*days
Arm/Group | Placebo + FOLFOX | Lidocaine + FOLFOX
Number analyzed (Participants) | 12 | 12
score on a scale*days
  pain AUC | 16.4 (18.3) | 9.5 (14.4)
  unpleasantness AUC | 33.1 (27.8) | 25.4 (22.6)
Statistical Analysis 1: Comparison: Placebo + FOLFOX vs Lidocaine + FOLFOX; Null hypothesis: Average AUC of cold pain score over 14 days of a chemotherapy cycle in the Control group is equal or lower than that of the experimental group. The comparison is for average AUC values over 7 cycles of chemotherapy per patient; Test type: Superiority; p = 0.318, t-test, 2 sided — p-value was not adjusted for any parameter; Mean Difference (Final Values) = 6.88, 95% CI 2-sided [-7.09 to 20.85]
Statistical Analysis 2: Comparison: Placebo + FOLFOX vs Lidocaine + FOLFOX; Null hypothesis: Cold hypersensitivity counted as unpleasantness score for 14 days after cycle (AUC) in the Control group is less than that of the experimental group. The difference was calculated for the Cycle 6 visit; Test type: Superiority; p = 0.466, t-test, 2 sided — p-value was not adjusted for any parameter; Mean Difference (Final Values) = 7.67, 95% CI 2-sided [-13.76 to 29.10]

2. Secondary Outcome: CIPN Score on EORTC QLQ-CIPN20
Description: Change in CIPN (Chemotherapy-induced peripheral Neuropathy) score (on EORTC QLQ-CIPN20 tool ) from baseline to the Cycle 6 (12 weeks), and from baseline to last follow-up (34-36 weeks). EORTC QLQ-CIPN20 ranges from 0 (no symptoms) to 100 (worst symptoms). A higher score represents worse neuropathy. The changes in scores are compared between study arms.
  EORTC QLQ-CIPN20 tool is a quality of life questionnaire (QLQ) from the European Organization for Research and Treatment of Cancer (EORTC) for evaluation of CIPN.
Time Frame: 12 weeks and 34-36 weeks
Population: Patients in each group who had corresponding visit data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo + FOLFOX | Lidocaine + FOLFOX
Number analyzed (Participants) | 12 | 12
score on a scale
  12 | 2 [0 to 8.3] | 4 [0 to 4]
  34-36 weeks | 17.0 [5.5 to 39.8] | 37.0 [7.4 to 47.2]
Statistical Analysis 1: Comparison: Placebo + FOLFOX vs Lidocaine + FOLFOX; the null hypothesis is EORTC QLQ-CIPN20 sensory score change in the Control group is equal to or less than that of the experimental group for the last follow-up study visit; Test type: Superiority; p = 0.338, Wilcoxon (Mann-Whitney) — p-value was not adjusted for any parameter; Median Difference (Final Values) = 20
Statistical Analysis 2: Comparison: Placebo + FOLFOX vs Lidocaine + FOLFOX; The null hypothesis is EORTC QLQ-CIPN20 sensory score change in the Control group is equal to or less than that of the experimental group for the cycle 6 (12 weeks) follow-up study visit; Test type: Superiority; p = 0.759, Wilcoxon (Mann-Whitney) — p-value was not adjusted for any parameter; Median Difference (Final Values) = 2

3. Secondary Outcome: Changes in NPSI Score.
Description: Changes in Neuropathic Pain Symptom Inventory (NPSI) descriptors of neuropathic pain over time from baseline to cycle 3(6 weeks), cycle 6 (12 weeks), and the last follow-up (34-36 weeks). The total NPSI score ranges from 0 to 100; a higher NPSI total score represents a worse neuropathy outcome. The changes in scores from baseline are compared between study arms.
Time Frame: 6 weeks, 12 weeks, 34-36 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo + FOLFOX | Lidocaine + FOLFOX
Number analyzed (Participants) | 12 | 12
score on a scale
  6 weeks visit | 0 [0 to 0] | 0 [0 to 0]
  12 weeks visit | 0 [0 to 0] | 0 [0 to 0]
  last follow-up visit | 3.0 [0.8 to 7.3] | 13.5 [0 to 17.3]
Statistical Analysis 1: Comparison: Placebo + FOLFOX vs Lidocaine + FOLFOX; The null hypothesis is NPSI total score in the Control group is equal to or less than that of the experimental group for the C3 (6 weeks) study visit; Test type: Superiority; p = 0.581, Wilcoxon (Mann-Whitney) — p-value was not adjusted for any parameter; Median Difference (Final Values) = 0
Statistical Analysis 2: Comparison: Placebo + FOLFOX vs Lidocaine + FOLFOX; The null hypothesis is NPSI total score in the Control group is equal to or less than that of the experimental group for the C6 (12 weeks) study visit; Test type: Superiority; p = 0.962, Wilcoxon (Mann-Whitney) — p-value was not adjusted for any parameter; Median Difference (Final Values) = 0
Statistical Analysis 3: Comparison: Placebo + FOLFOX vs Lidocaine + FOLFOX; The null hypothesis is NPSI total score in the Control group is equal to or less than that of the experimental group for the last follow-up study visit; Test type: Superiority; p = 0.365, Wilcoxon (Mann-Whitney) — p-value was not adjusted for any parameter; Median Difference (Final Values) = 10.50

4. Secondary Outcome: The Cumulative Dose of Oxaliplatin
Description: The cumulative dose of oxaliplatin received over the course (up to 12 cycles) of mFOLFOX6 treatment regimen. It corresponds to the absolute summed up quantity of Oxaliplatin administered to the patient over time. There is no range for this measure. Since this is a dose-limiting neuropathy prevention study, the higher value can be interpreted as better outcome.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo + FOLFOX | Lidocaine + FOLFOX
Number analyzed (Participants) | 12 | 12
mg | 1161.8 (300.2) | 1294.8 (221.6)
Statistical Analysis 1: Comparison: Placebo + FOLFOX vs Lidocaine + FOLFOX; The null hypothesis is Oxaliplatin cumulative dose in the Control group is equal to or higher than that of the experimental group; Test type: Superiority; p = 0.730, t-test, 2 sided; Mean Difference (Final Values) = 57.68, 95% CI 2-sided [-1771 to 1886]

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse Event: any unfavorable medical occurrence in a human subject including any abnormal sign, symptom, or disease.
  For the purposes of this protocol, all adverse events will be collected and documented on CRFs by questionnaire.
Arm/Group | Placebo + FOLFOX | Lidocaine + FOLFOX
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 6/12 | 12/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + FOLFOX (N=12) | Lidocaine + FOLFOX (N=14)
Dizziness (Nervous system disorders) | 4 (14) | 4 (14)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (5)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 6 (12)
Lightheadedness (Nervous system disorders) | 1 (1) | 2 (4)
Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, the study finished earlier than planned. The total number of patients enrolled was 26 instead of 30.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03254394/Prot_SAP_000.pdf